CLINICAL TRIAL: NCT01990326
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled Study of XAF5 Gel for Reduction of Submental Fat
Brief Title: Safety and Feasibility Study of XAF5 Gel for Reduction of Submental Fat
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Feasibility cohorts competed. Efficacy cohort not initiated for business reasons
Sponsor: Topokine Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XAF5 B1
Record Dates: First submitted 2013-11-01; First posted 2013-11-21 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2014-07

CONDITIONS: Excess Submental Fat ("Double Chin")

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XAF5 Gel (Experimental): The patient will apply XAF5 Gel to the skin of the submental area once a night.
  Interventions: Drug: XAF5 Gel
- Placebo Gel (Placebo Comparator): The patient will apply a Placebo Gel to the skin of the submental area once a night.
  Interventions: Drug: Placebo Gel

INTERVENTIONS:
Drug: XAF5 Gel
  Arms: XAF5 Gel
Drug: Placebo Gel
  Arms: Placebo Gel

SUMMARY:
This study will test the effects of XAF5 Gel (applied to skin each night for 6 weeks) on excess submental fat, also known as double chin. The study will also assess the safety and tolerability of XAF5 Gel.

ELIGIBILITY:
Inclusion Criteria (paraphrased):

* Adult men and women
* Must understand and provide informed consent
* Moderate submental fat (as determined by the clinician)
* No laxity (looseness) or minimal laxity of submental skin
* Healthy skin upon which a skin reaction would be visible

Exclusion Criteria (paraphrased):

* A clinically significant health problem or recent illness
* A clinically significant abnormal result on physical exam or laboratory tests
* Neck or facial hair that would interfere with applying the study drug to submental skin
* Clinically significant skin disease
* Body Mass Index (BMI) >= 40
* Plan to begin a diet or weight loss regimen during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events | From Day 1 to Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Singer, M.D., Ph.D., Study Director — Topokine Therapeutics